CLINICAL TRIAL: NCT00338598
Title: Facilitation of NMDA Receptor Function in Patients With Schizophrenia and Co-morbid Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20915
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Alcoholism; Schizophrenia
Keywords: glycine; treatment; alcohol dependence; schizophrenia
MeSH Terms: conditions — Alcoholism; Schizophrenia | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycine (Experimental): Glycine, 0.8 gr per kg given in two daily doses
  Interventions: Drug: Glycine
- placebo (Placebo Comparator): placebo will be administered.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Glycine — Glycine, 0.8 gr per kg given in two daily doses
  Arms: Glycine
Drug: placebo
  Arms: placebo

SUMMARY:
This placebo-controlled study is designed to evaluate the efficacy of glycine, an agonist of the glycine-B co-agonist site of the NMDA receptor, on alcohol consumption and craving as well as negative symptoms in schizophrenia.

Glycine will decrease the rewarding action of ethanol and reduce ethanol consumption. Also, glycine will improve negative symptoms and cognitive deficits in schizophrenia.

DETAILED DESCRIPTION:
OBJECTIVE: Schizophrenia affects about 1% of the general population and is a highly disabling disease. Additionally, the rate of alcohol dependency for patients with schizophrenia is very high. There are no established treatments for alcohol dependency and negative symptoms in schizophrenia. This study will examine whether the addition of glycine to neuroleptic medications will help patients with schizophrenia and alcoholism decrease their drinking as well as improve negative symptoms.

RESEARCH PLAN: An abnormality of the glutamate neurotransmitter system has been hypothesized for both alcoholism and schizophrenia. Studies suggest that the amino acid glycine may improve alcohol dependency and symptoms of schizophrenia by acting on the N methyl D aspartate (NMDA) glutamate receptor. Glycine causes reversal of the effects of ethanol in animal studies and improves mood, social withdrawal and other so called "negative symptoms" of schizophrenia. Consequently, the use of glycine by patients with schizophrenia and alcohol dependency may potentially decrease alcohol craving and alcohol consumption and also improve certain symptoms of schizophrenia. The potential of glycine to improve both alcohol dependency and negative symptoms could represent an important step in the improvement of the quality of life for patients with schizophrenia.

METHODOLOGY/FINDINGS/RESULTS: In order to test this hypothesis, we will use a double blind, placebo controlled study and measure the number of drinks, the degree of craving for alcohol and symptoms of schizophrenia among other parameters. Our principal approach to analyses of medication effectiveness will be the application of the linear mixed effect model. The linear mixed effect model permits a flexible approach for studying change in individuals through time as a random effect, and does not require all patients to have data at all measured points. Our principal model of analysis includes treatment (placebo or glycine), as between subject factor, and time, as within subject factor. Compliance will be also included as a time varying independent variable. This project continues to recruit subjects.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* DSM-IV diagnosis of alcohol dependence
* Stable treatment with typical or atypical antipsychotics

Exclusion Criteria:

* Axis I diagnosis other than alcohol dependence, schizophrenia, schizoaffective disorder, OCD, and PTSD.
* current drug dependence
* evidence of significant hepatocellular injury evidence by abnormal SGOT or SGPT levels
* history of seizures
* diabetes and medical conditions that would alter glycine metabolism
* positive pregnancy test
* treatment with clozapine, naltrexone or disulfiram

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the VA hospital in West Haven, CT and the Community Mental Health Center in New Haven, CT through word of mouth, advertisement and clinician referrals.
Pre-assignment Details: Twenty men, who met DSM IV criteria for schizophrenia or schizoaffective disorder, who also met DSM IV diagnosis of alcohol dependence with at least one recent episode of heavy drinking (defined as more than 5 drinks/drinking episode) over the past 14 days participated in the study. The participants were in stable treatment for at least 2 weeks.
Groups:
- Placebo: placebo will be administered.
  placebo
Period: Overall Study
Arm/Group | Glycine | Placebo
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycine | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (4.8) | 48.6 (5.0) | 48.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 2 | 9
  Black | 3 | 7 | 10
Drinks per day [Mean (Standard Deviation); unit: drinks per day] | 8.9 (8.5) | 5.9 (5.0) | 7.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Weekly Alcohol Consumption
Description: Percentage of drinking days and heavy drinking days using timeline follow back
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 10 | 10
percentage of days
  % number of drinking days | 23.4 (28.8) | 19.6 (29.0)
  % number of heavy drinking days | 15.7 (20.8) | 10.0 (12.6)

2. Primary Outcome: Self Reported Weekly Alcohol Craving
Description: The Obsessive Compulsive Drinking Scale (OCDS) is consisted by 14 items rated 0 - 4. The minimum and maximum values possibly obtained in this scale are respectively 0 and 56, this last one, meaning the most craving possible experienced. It is a short and easy to administer scale (average of 5 minutes per self-rating), built to measure severity and improvement during alcoholism treatment trials.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 16.1 (3.1) | 17.5 (3.2)
  Week 12 | 10.2 (3.1) | 12.1 (3.3)

3. Primary Outcome: Weekly Ratings of Negative/Positive Psychotic Symptoms
Description: The PANSS or the Positive and Negative Syndrome Scale is a medical scale used for measuring symptom severity of patients with schizophrenia. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale.The scores for these scales are arrived at by summation of ratings across component items. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. A higher score indicates more severe symptoms for each scale.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline Positive | 16.3 (1.3) | 15.3 (1.3)
  Week 12 Positive | 12.0 (1.3) | 13.5 (1.4)
  Baseline Negative | 16.7 (1.5) | 12.5 (1.6)
  Week 12 Negative | 14.9 (1.5) | 13.0 (1.6)
  Baseline General | 32.4 (2.5) | 29.4 (2.6)
  Week 12 General | 31.9 (2.5) | 29.8 (2.7)

4. Primary Outcome: Baseline and End of Treatment Cognitive Functioning Measures (Hopkins)
Description: Hopkins Verbal Learning Test Assesses short term verbal learning and memory. Subscales include immediate recall (0-36), delayed recall (0-12) , and recognition (0-12). A higher score indicates better memory performance.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline Immediate Recall | 21.8 (1.7) | 19.7 (1.7)
  12 Weeks Immediate Recall | 20.9 (1.8) | 19.5 (1.8)
  Baseline Delayed Recall | 6.1 (0.9) | 6.4 (0.9)
  12 Weeks Delayed Recall | 6.6 (0.9) | 6.5 (0.9)
  Baseline Recognition | 10.2 (1.0) | 12.5 (1.0)
  12 Weeks Recognition | 9.8 (1.0) | 12.2 (1.0)

5. Secondary Outcome: Weekly Drug Use
Time Frame: 12 weeks
Population: Data was not collected
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Baseline and End of Treatment Quality of Life
Time Frame: 12 weeks
Population: Data was not collected
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Baseline and End of Treatment Neurophysiological Measures
Time Frame: 12 weeks
Population: Data was not collected
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Glycine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycine (N=10) | Placebo (N=10)
ER for intoxication (General disorders) | 0 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ER Visit (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Relapse (General disorders) | 1 | 0
auditory hallucinations (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes